CLINICAL TRIAL: NCT02370459
Title: Adolescent AFIX: A Multi-state RCT to Increase Adolescent Vaccination by Facilitating Providers' Adoption of Best Practices
Brief Title: AFIX to Improve HPV Vaccination
Acronym: AFIX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Robert Wood Johnson Foundation (Other); Washington State, Department of Health (Other Government); Illinois Department of Public Health (Other); Michigan Department of Community Health (Other); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 13-3599; 71272 (Other Grant/Funding Number: Robert Wood Johnson Foundation)
Record Dates: First submitted 2015-02-05; First posted 2015-02-25 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Papillomavirus Vaccines; Adolescent Health Services
Keywords: Papillomavirus Vaccines; Immunization; Quality Improvement; Adolescent Health Services
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- control (No Intervention): This arm includes 30 high-volume primary care clinics in each of three states (Washington, Illinois, Michigan) for a total of 90 clinics. Clinics randomly assigned to this arm will receive no AFIX consultation.
- AFIX in-person consultation (Experimental): This arm includes 30 high-volume primary care clinics in each of three states (Washington, Illinois, Michigan) for a total of 90 clinics. Clinics randomly assigned to this arm will receive an in-person AFIX consultation. Consultations will be delivered by state health department staff.
  Interventions: Other: AFIX in-person consultation
- AFIX webinar consultation (Experimental): This arm includes 30 high-volume primary care clinics in each of three states (Washington, Illinois, Michigan) for a total of 90. Clinics randomly assigned to this arm will receive an AFIX consultation via interactive webinar. Consultations will be delivered by state health department staff.
  Interventions: Other: AFIX webinar consultation

INTERVENTIONS:
Other: AFIX in-person consultation — The adolescent AFIX (Assessment, Feedback, Incentives, and eXchange) Program is a quality improvement strategy developed by the CDC to improve the immunization practices and vaccination coverage levels of public and private health care providers. It has four main components: 1) Assessment of a provider's current immunization practices and vaccination levels, 2) Feedback of the assessment results and strategies to improve coverage levels, 3) Incentives to improve coverage levels, and 4) eXchange of information and resources necessary to facilitate improvement. Relevant AFIX information will be communicated to vaccine providers using several intervention and quality improvement components.
  Other Names: AFIX, Assessment, Feedback, Incentives, and eXchange Program
  Arms: AFIX in-person consultation
Other: AFIX webinar consultation — The adolescent AFIX (Assessment, Feedback, Incentives, and eXchange) Program is a quality improvement strategy developed by the CDC to improve the immunization practices and vaccination coverage levels of public and private health care providers. It has four main components: 1) Assessment of a provider's current immunization practices and vaccination levels, 2) Feedback of the assessment results and strategies to improve coverage levels, 3) Incentives to improve coverage levels, and 4) eXchange of information and resources necessary to facilitate improvement. Relevant AFIX information will be communicated to vaccine providers using several intervention and quality improvement components.
  Other Names: AFIX, Assessment, Feedback, Incentives, and eXchange Program
  Arms: AFIX webinar consultation

SUMMARY:
The University of North Carolina will test the effectiveness of the Centers for Disease Control and Prevention's AFIX model for increasing HPV vaccination coverage among adolescents. AFIX (Assessment, Feedback, Incentives and eXchange) consists of brief quality improvement consultations that immunization specialists from state health departments deliver to vaccine providers in primary care settings. Using immunization registry data, the specialist evaluates the clinic's vaccination coverage and delivers education on best practices to improve coverage. We will compare changes in HPV vaccination coverage before and after consultations for high-volume pediatric and family medicine clinics across three study conditions: traditional consultations (in-person group), virtual consultations (webinar group), or no consultations (control group). In each participating state, 30 clinics will be randomly assigned to each study arm, for a total of 90 clinics per state, or 270 clinics overall. The primary objective of this study is to compare the change in coverage for HPV vaccine initiation among 11-12 year old patients, from baseline to 6-month follow-up. Secondarily, we will compare the change in coverage for other vaccines and age groups.

ELIGIBILITY:
Inclusion Criteria: Pediatric or family medicine clinics or practices in WA, IL, or MI with

* at least 500 active records for patients, ages 11-17, in their states' immunization information systems.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2015-04; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
HPV vaccination (≥1 dose), 11-12 year olds | Six months
  Coverage change from baseline to six months in HPV vaccine initiation (≥1 dose), among 11- to 12-year old patients in the control arm versus the combined in-person and webinar intervention arms, as measured by electronic immunization information system (IIS) records, controlling for child's sex

SECONDARY OUTCOMES:
HPV vaccination (≥1 dose), 11-12 year olds | Six months
  Coverage change from baseline to six months in HPV vaccine initiation (≥1 dose), among 11- 12-year old patients in the control arm versus the combined in-person and webinar intervention arms, as measured by IIS records, stratifying by child's sex.
HPV vaccination (≥1 dose), 11-12 year olds | Six months
  Coverage change from baseline to six months in HPV vaccine initiation (≥1 dose), among 11- to 12-year-old patients in the control arm versus the combined in-person and webinar intervention arms, as measured by IIS records, stratifying by state (IL, MI or WA).
HPV vaccination (≥1 dose), 11-12 year olds | Twelve months
  Coverage change from baseline to twelve months in HPV vaccine initiation (≥1 dose), among 11- to 12-year-old patients in the control arm versus the combined in-person and webinar intervention arms, as measured by IIS records, stratifying by child's sex.
HPV vaccination (≥1 dose), 11-12 year olds | Twelve months
  Coverage change from baseline to twelve months in HPV vaccine initiation (≥1 dose), among 11- to 12-year-old patients in the control arm versus the combined in-person and webinar intervention arms, as measured by IIS records, stratifying by state (IL, MI or WA).
HPV vaccination (3 doses), 11-12 year olds | Six months
  Coverage change from baseline to six months in HPV vaccine completion (3 doses), among 11- to 12-year-old patients in the control arm versus the combined in-person and webinar intervention arms, as measured by IIS records.
Tetanus, diphtheria, and acellular pertussis (Tdap) vaccination, 11-12 year olds | Six months
  Coverage change from baseline to six months in Tdap vaccination among 11- to 12-year-old patients in the control arm versus the combined in-person and webinar intervention arms, as measured by IIS records.
Meningococcal vaccination (≥1 dose), 11-12 year olds | Six months
  Coverage change from baseline to six months in meningococcal vaccination (≥1 dose), among 11- to 12-year-old patients in the control arm versus the combined in-person and webinar intervention arms, as measured by IIS records.
HPV vaccination (≥1 dose), 13-17 year olds | Six months
  Coverage change from baseline to six months in HPV vaccine initiation (≥1 dose), among 13- to 17-year-old patients in the control arm versus the combined in-person and webinar intervention arms, as measured by IIS records.
HPV vaccination (3 doses), 13-17 year olds | Six months
  Coverage change from baseline to six months in HPV vaccine completion (3 doses), among 13- to 17-year-old patients in the control arm versus the combined in-person and webinar intervention arms, as measured by IIS records.
Tdap vaccination, 13-17 year olds | Six months
  Coverage change from baseline to six months in Tdap vaccination among 13- to 17-year-old patients in the control arm versus the combined in-person and webinar intervention arms, as measured by IIS records.
Meningococcal vaccination (≥1 dose), 13-17 year olds | Six months
  Coverage change from baseline to six months in meningococcal vaccination (≥1 dose), among 13- to 17-year-old patients in the control arm versus the combined in-person and webinar intervention arms, as measured by IIS records.
HPV vaccination (≥1 dose), 11-12 year olds | Twelve months
  Coverage change from baseline to twelve months in HPV vaccine initiation (≥1 dose), among 11- to 12-year-old patients in the control arm versus the combined in-person and webinar intervention arms, as measured by IIS records.
HPV vaccination (3 doses), 11-12 year olds | Twelve months
  Coverage change from baseline to twelve months in HPV vaccine completion (3 doses), among 11- to 12-year-old patients in the control arm versus the combined in-person and webinar intervention arms, as measured by IIS records.
Tdap vaccination, 11-12 year olds | Twelve months
  Coverage change from baseline to twelve months in Tdap vaccination among 11- to 12-year-old patients in the control arm versus the combined in-person and webinar intervention arms, as measured by IIS records.
Meningococcal vaccination (≥1 dose), 11-12 year olds | Twelve months
  Coverage change from baseline to twelve months in meningococcal vaccination (≥1 dose), among 11- to 12-year-old patients in the control arm versus the combined in-person and webinar intervention arms, as measured by IIS records.
HPV vaccination (≥1 dose), 13-17 year olds | Twelve months
  Coverage change from baseline to twelve months in HPV vaccine initiation (≥1 dose), among 13- to 17-year-old patients in the control arm versus the combined in-person and webinar intervention arms, as measured by IIS records.
HPV vaccination (3 doses), 13-17 year olds | Twelve months
  Coverage change from baseline to twelve months in HPV vaccine completion (3 doses), among 13- to 17-year-old patients in the control arm versus the combined in-person and webinar intervention arms, as measured by IIS records.
Tdap vaccination, 13-17 year olds | Twelve months
  Coverage change from baseline to twelve months in Tdap vaccination among 13- to 17-year-old patients in the control arm versus the combined in-person and webinar intervention arms, as measured by IIS records.
Meningococcal vaccination (≥1 dose), 13-17 year olds | Twelve months
  Coverage change from baseline to twelve months in meningococcal vaccination (≥1 dose), among 13- to 17-year-old patients in the control arm versus the combined in-person and webinar intervention arms, as measured by IIS records.
HPV vaccination (≥1 dose), 11-12 year olds | Six months
  Coverage change from baseline to six months in HPV vaccine initiation (≥1 dose), among 11- to 12-year-old patients in the webinar versus in-person intervention arm, as measured by IIS records.
HPV vaccination (3 doses), 11-12 year olds | Six months
  Coverage change from baseline to six months in HPV vaccine completion (3 doses), among 11- to 12-year-old patients in the webinar versus in-person intervention arm, as measured by IIS records.
Tdap vaccination, 11-12 year olds | Six months
  Coverage change from baseline to six months in Tdap vaccination among 11- to 12-year-old patients in the webinar versus in-person intervention arm, as measured by IIS records.
Meningococcal vaccination (≥1 dose), 11-12 year olds | Six months
  Coverage change from baseline to six months in meningococcal vaccination (≥1 dose), among 11- to 12-year-old patients in the webinar versus in-person intervention arm, as measured by IIS records.
HPV vaccination (≥1 dose), 13-17 year olds | Six months
  Coverage change from baseline to six months in HPV vaccine initiation (≥1 dose), among 13- to 17-year-old patients in the webinar versus in-person intervention arm, as measured by IIS records.
HPV vaccination (3 doses), 13-17 year olds | Six months
  Coverage change from baseline to six months in HPV vaccine completion (3 doses), among 13- to 17-year-old patients in the webinar versus in-person intervention arm, as measured by IIS records.
Tdap vaccination, 13-17 year olds | Six months
  Coverage change from baseline to six months in Tdap vaccination among 13- to 17-year-old patients in the webinar versus in-person intervention arm, as measured by IIS records.
Meningococcal vaccination (≥1 dose), 13-17 year olds | Six months
  Coverage change from baseline to six months in meningococcal vaccination (≥1 dose), among 13- to 17-year-old patients in the webinar versus in-person intervention arm, as measured by IIS records.
HPV vaccination (≥1 dose), 11-12 year olds | Twelve months
  Coverage change from baseline to twelve months in HPV vaccine initiation (≥1 dose), among 11- to 12-year-old patients in the webinar versus in-person intervention arm, as measured by IIS records.
HPV vaccination (3 doses), 11-12 year olds | Twelve months
  Coverage change from baseline to twelve months in HPV vaccine completion (3 doses), among 11- to 12-year-old patients in the webinar versus in-person intervention arm, as measured by IIS records.
Tdap vaccination, 11-12 year olds | Twelve months
  Coverage change from baseline to twelve months in Tdap vaccination among 11- to 12-year-old patients in the webinar versus in-person intervention arm, as measured by IIS records.
Meningococcal vaccination (≥1 dose), 11-12 year olds | Twelve months
  Coverage change from baseline to twelve months in meningococcal vaccination (≥1 dose), among 11- to 12-year-old patients in the webinar versus in-person intervention arm, as measured by IIS records.
HPV vaccination (≥1 dose), 13-17 year olds | Twelve months
  Coverage change from baseline to twelve months in HPV vaccine initiation (≥1 dose), among 13- to 17-year-old patients in the webinar versus in-person intervention arm, as measured by IIS records.
HPV vaccination (3 doses), 13-17 year olds | Twelve months
  Coverage change from baseline to twelve months in HPV vaccine completion (3 doses), among 13- to 17-year-old patients in the webinar versus in-person intervention arm, as measured by IIS records.
Tdap vaccination, 13-17 year olds | Twelve months
  Coverage change from baseline to twelve months in Tdap vaccination among 13- to 17-year-old patients in the webinar versus in-person intervention arm, as measured by IIS records.
Meningococcal vaccination (≥1 dose), 13-17 year olds | Twelve months
  Coverage change from baseline to twelve months in meningococcal vaccination (≥1 dose), among 13- to 17-year-old patients in the webinar versus in-person intervention arm, as measured by IIS records.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa B Gilkey, PhD, Principal Investigator — Harvard Medical School (HMS and HSDM); Noel T Brewer, PhD, Principal Investigator — University of North Carolina
Locations (4):
- United States (4):
  - Illinois Department of Public Health, Springfield, Illinois
  - Michigan Department of Community Health, Lansing, Michigan
  - University of North Carolina, Chapel Hill, North Carolina
  - Washington State Department of Health, Olympia, Washington

IPD SHARING:
Plan to Share IPD: No
No raw data will be shared with the general public or other researchers.